CLINICAL TRIAL: NCT02856763
Title: Predictive Factors of ANTI-TNF Response in Luminal Crohn's Disease Complicated by Abscess A Multicenter Prospective, Observational Cohort Study
Brief Title: Predictive Factors of ANTI-TNF Response in Luminal Crohn's Disease Complicated by Abscess
Acronym: MICA
Status: Completed | Type: Observational
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Other Study IDs: GETAID 2012-1; 2012-000982-19 (EudraCT Number)
Record Dates: First submitted 2015-06-21; First posted 2016-08-05 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: CD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To identify predictive factors of adalimumab (anti TNF) response in patients with luminal Crohn's disease complicated by intra-abdominal and/or pelvic abscess after complete resolution of infection.

DETAILED DESCRIPTION:
Multicenter prospective observational cohort.

Initial management of sepsis and abscess (Before anti-TNF therapy initiation) i. Antibiotics. ii. Percutaneous drainage will be performed every time when possible iii. Surgical drainage will be performed if percutaneous drainage is not accessible or fails iv.

Concomitant medications :

* Steroids will be rapidly tapered and stopped.
* Azathioprine, 6-mercaptopurtine, 5-ASA derivatives and methotrexate will be maintained at a stable dose.
* If not present at inclusion, immunosuppressors could be introduced at the discretion of investigator
* Antibiotics could be used if needed for infections not related to intra-abdominal abscess recurrence and Crohn's disease. v.

Supportive care including artificial nutrition will be started if necessary.

2. Anti-TNF therapy:

- The anti-TNF agent will be adalimumab, administered as subcutaneous injection of 160 mg at W0, 80 mg at W2, followed by 40 mg every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years.
* Diagnosis of Crohn's disease (confirmed by clinical evaluation and a combination of endoscopic, histological, radiological, and/or biochemical investigations according to European guidelines)
* AND diagnosis of spontaneous intra-abdominal and/or pelvic abscess according to radiologic criteria confirmed by US, CT or magnetic resonance enterography (MRE).
* In patients who have not responded despite a full and adequate course of therapy with a corticosteroid and/or an immunosuppressant or who are intolerant to or have medical contraindications for such therapies
* Written consent MAIN

Exclusion Criteria:

* Age under 18 years. - Absence of written consent. - Post-operative abscess (occurring within 12 weeks after intestinal resection). - Isolated intra-parietal abscess of small intestine or colon. - Need for immediate surgery including irreversible bowel obstruction, peritonitis or uncontrolled sepsis. - Perineal abscess complicating perianal Crohn's disease. - Abscess developing under anti-TNF therapy. - Previous failure or intolerance to adalimumab. - Contraindication to anti-TNF therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting a luminal Crohn's disease complicated by an intra abdominal and/or pelvic abscess meeting the inclusion criteria and followed or addressed in one of the participating centers will be enrolled in the pre-inclusion phase of the study consisting in abscess drainage and antibiotic therapy as recommended by local and European guidelines.
  - After the initial pre-inclusion phase of the study, if there is a complete resolution of sepsis and abscess confirmed by MRE, patients for whom the treating physician decides to introduce adalimumab according to local and European Guidelines will be included in the anti-TNF treatment phase.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Identification of predictive factors of adalimumab (anti TNF) failure at Week 24. | Week 24
  W24 adalimumab failure in this context is defined as: o Need for intestinal resection, o or Need to begin steroids after 12 weeks of adalimumab treatment, o or Abscess recurrence confirmed by MRE, o or Clinical relapse defined as CDAI > 220 or HBI > 4 (table 3) and CRP > 10 mg/L at two consecutive visits

SECONDARY OUTCOMES:
Clinical Remission | Week 48
  - Clinical remission (CDAI <150 or HBI ≤ 4) at each visit until W48
Monitoring of obstructive symptoms | Week 48
  - Monitoring of obstructive symptoms to determine the degree of CD related bowel obstruction (Obstructive abdominal pain, nausea, vomiting, dietary restriction due to symptoms, bowel obstruction, cf. table 3) at each visit until W48.
Evolution of items measured by MRE | Week 24
  Evolution of items measured by MRE between inclusion and week 24
hospital stay | Week 48
  - Length of hospital stay.
SAE | Week 48
  - Serious adverse events or severe infections leading to definitive treatment withdrawal.
Death | Week 24
  Death related to CD between D0 and W24.

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Bouhnik, MD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Guillaume Pineton de Chambrun, MD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (2):
- France (2):
  - Beaujon Hospital, Clichy
  - Aphp St Louis, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bouhnik Y, Pineton de Chambrun G, Lambert J, Nachury M, Seksik P, Altwegg R, Vuitton L, Stefanescu C, Nancey S, Aubourg A, Serrero M, Filippi J, Desseaux K, Viennot S, Abitbol V, Boualit M, Bourreille A, Giletta C, Buisson A, Roblin X, Dib N, Malamut G, Amiot A, Fumery M, Louis E, Elgharabawy Y, Peyrin-Biroulet L; MICA-GETAID Study Group. Adalimumab in Biologic-naive Patients With Crohn's Disease After Resolution of an Intra-abdominal Abscess: A Prospective Study From the GETAID. Clin Gastroenterol Hepatol. 2023 Dec;21(13):3365-3378.e5. doi: 10.1016/j.cgh.2023.01.013. Epub 2023 Jan 31. PMID 36731588